CLINICAL TRIAL: NCT03275194
Title: Hyperthermic Intraperitoneal Chemotherapy in Ovarian Carcinoma Clinical Stage IIIC and IV During Interval Laparotomy. Phase II Study
Brief Title: HIPEC in Ovarian Carcinoma Clinical Stage IIIC and IV During Interval Laparotomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Rosa A. Salcedo, Surgical oncologist, Gynecology oncology division, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INCAN/CI/483/15
Record Dates: First submitted 2017-09-02; First posted 2017-09-07 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: HPEC; Ovarian Cancer; Women's Health: Neoplasm of Ovary; Chemotherapy Effect
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data will be evaluated for a external person with the groups labeled as "A" and "B" for all outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): After achieving a complete cytoreductive surgery (no visible residual disease), the patient will be randomised and if is assigned to this arm does not receive additional treatment and the procedure will be finished.
- HIPEC group (Experimental): After achieving a complete cytoreductive surgery (no visible residual disease), the patient will be randomised and if is assigned to this arm receive a HIPEC procedure with cisplatin and doxorubicin.
  Interventions: Procedure: HIPEC

INTERVENTIONS:
Procedure: HIPEC — Following complete cytoreductive surgery without any evidence of residual disease, the patient will be randomized either HIPEC (intervention) or no-HIPEC (control) in the operative Room. If the arm HIPEC is obtained, then a HIPEC procedure with cisplatin and doxorubicin will be performed. If no-HIPEC (control arm) is assigned then the surgical procedure will be finished.
  Arms: HIPEC group

SUMMARY:
Ovarian cancer is the leading cause of gynecological cancer mortality, with no current screening method effective for early diagnosis, with 75% of advanced stage patients being detected. Not all patients are candidates for standard treatment, which is primary cytoreduction followed by adjuvant chemotherapy, due to the advanced process. A subgroup of patients will receive neoadjuvant chemotherapy followed by interval surgery, which allows higher rates of optimal cytoreduction with low morbidity and mortality. Hyperthermic intraperitoneal chemotherapy (HIPEC) is a therapeutic option that is used in pathologies of peritoneal dissemination, whose morbidity and mortality has been reported in several series and is promising as a management option for ovarian cancer, so it is necessary to evaluate morbidity and mortality that conditions this modality of treatment as well as if it impacts on the quality of life of the patients to whom they are performed, which will allow offering our patients an option of additional treatment to the standard.

DETAILED DESCRIPTION:
Ovarian cancer ranks seventh in incidence of malignant neoplasms in women younger than 65 years and is the leading cause of cancer death in women in the United States. Due to the absence of an effective screening method and early symptoms, 70% of the cases are diagnosed in advanced clinical stage (stage III or IV) and the overall 5-year survival is 30-40%.

The standard treatment of locally advanced ovarian carcinoma is primary cytoreductive surgery plus adjuvant chemotherapy with carboplatin and taxanes. In cases where it is not possible to perform primary cytoreductive surgery a treatment option is to start with induction chemotherapy (three or four cycles), in order to reduce tumor size and volume, after which it is performed an interval surgery, during which it has been reported that optimal cytoreduction is achieved in 77-94% of patients, with lower morbidity and mortality than primary surgery, without oncological compromise. Subsequent to interval surgery three additional cycles of chemotherapy are applied.

Despite an adequate response to the treatment aforementioned, 70% of patients will recur within the first two years. Because of this high recurrence rate, other therapeutic alternatives have been evaluated, among them is hyperthermic intraperitoneal chemotherapy (HIPEC). Since its first description 20 years ago, the HIPEC associated with cytoreductive surgery in the treatment of malignant neoplasms (primary or metastatic) in the peritoneal surface has become the standard of treatment, specifically in patients with peritoneal pseudomyxoma, peritoneal mesothelioma, and cancer with limited peritoneal involvement. In ovarian cancer, attempts are being made to determine its usefulness in specific scenarios of this disease.

The increasing interest in the use of HIPEC in the management of advanced ovarian cancer is based on the coelomic dissemination of ovarian cancer, which in theory would allow this modality of treatment to be effective. Moreover, optimal cytoreduction and administration of intraperitoneal chemotherapy over intravenous (intraperitoneal normothermy) have been shown to be superior in achieving higher survival rates in randomised trials.

Few groups in the world have studied the use of HIPEC in ovarian cancer, however, studies have been (and are being conducted) in the following scenarios: a) during primary cytoreduction, b) during interval laparotomy, c) as consolidation after standard treatment, d) recurrence of platinum resistant carcinoma and e) in the recurrence of "platinum sensitive" carcinoma. The morbidity of this procedure reported in different series is 33-39%, and mortality of 0-9%. The feasibility of the procedure with low rates of morbidity and mortality has been reported, specially when the treatment is done by a multidisciplinary group especially trained in HIPEC.

The present project is a Phase II, randomised study whose primary objective is to evaluate the morbidity, mortality, and quality of life of patients undergoing HIPEC during the surgery with optimal surgical cytoreduction. One group will be treated with cytoreduction and adjuvant chemotherapy, while the experimental group will be treated with cytoreduction followed by HIPEC. Our secondary objectives are the assessment of the disease-free period and overall survival. The working hypothesis is that the use of HIPEC during interval surgery will have a morbidity considered as acceptable as reported in the literature without significant deterioration in the quality of life.

The importance of evaluating this new therapeutic tool is that any of the current treatments for ovarian cancer have a high rate of recurrence. Based in the evidence, biological behaviour and pattern of dissemination of ovarian cancer, treatment should incorporate both systemic and locoregional therapy, because the neoplasm spreads via coelomic, lymphatic and hematogenous. The use of HIPEC together with the surgical event of cytoreduction could avoid recurrence and allow us to distinguish those patients who are candidates for this procedure and their actual benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients younger than 70 years
2. Patient with a diagnosis of high grade serous carcinoma of the ovary and low-grade endometrioid corroborated by histopathological study.
3. Clinical stage IIIC and IVA (cytology-positive pleural effusion) who have received induction chemotherapy 3 or 4 cycles of CARBOPLATIN and PACLITAXEL.
4. Partial response to treatment with chemotherapy and evaluated by computed tomography (RECIST-see below) and response of at least 50% by serum determination of CA-125 antigen.
5. Signature of informed consent.
6. Optimal cytoreduction with residual tumor less than 2.5 mm during interval surgery
7. ECOG less than or equal to 1
8. Adequate renal, cardiac, hepatic, bone marrow and lung function evaluated preoperatively with the following parameters:

   a) Hb equal to or greater than 10 g / L (pre-treatment transfusion is permitted to achieve this hemoglobin level) b) Leukocytes Greater than 3000 / mm3 (c) Platelets equal to or greater than 100 000 / mm3 (d) total bilirubin less than 1.5 times greater than the normal value e) Hepatic transaminases less than 1.5 times higher than normal value f) Creatinine <1.2 g / dl. In case of being elevated the measured purification should be greater than 60mL / min according to Cockroft's formula.

   g) Albumin greater than 3gr / dl. h) Left Ventricle Ejection fraction per cardiac echography greater than 55% 9). Sugarbaker carcinomatosis index less than 20

Exclusion Criteria:

1. Patients with heart failure, ischemic heart disease
2. Previous history of treatment with chemotherapy for some other neoplasia
3. History of neuropsychiatric disease
4. Patients with intra operative bleeding that condition hemodynamic instability.
5. Patient requiring more than 2 intraoperative anastomosis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Genotypic sex
Enrollment: 100 (Estimated)
Dates: Start 2017-09-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 1 year
  To assess the mortality associated with the use of intraperitoneal hyperthermic chemotherapy during interval laparotomy.
Impact of quality of life | Up to 1 year
  To evaluate the impact on patients' quality of life, which is undergoing intraperitoneal hyperthermic chemotherapy during interval laparotomy. The scales that will be used will be EORTC QLQ-C30 (Ver. 3) and EORTC QLQ-OV28.
Morbility | Up to 1 year
  To assess the morbidity associated with the use of intraperitoneal hyperthermic chemotherapy during interval laparotomy.

SECONDARY OUTCOMES:
Disease free survival | Up to 2 years
  Evaluate disease-free survival.
Overall survival | up to five years
  Evaluate overall 5 year survival.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa A Salcedo-Hernandez, MSc, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The database without any patient identity data could be accede for anyone asking for.